CLINICAL TRIAL: NCT05416268
Title: An Objective Study to Compare the Diopsys NOVA and LKC RETeval Devices Using the Diopsys LID Electrodes and the LKC RETeval Self-Adhering Electrode Arrays
Brief Title: Study to Compare the Diopsys NOVA and LKC RETeval Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diopsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 200
Record Dates: First submitted 2022-06-01; First posted 2022-06-13 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases | interventions — Electroretinography

STUDY DESIGN:
Intervention Model Description: This study is an open label, prospective study comparing the Diopsys NOVA and LKC RETeval devices using the Diopsys Lid Electrodes and the LKC RETeval Self-Adhering Electrode Arrays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Diopsys NOVA and Diopsys Electrodes (Other): Subjects will receive the PhNR test three times using the Diopsys device and Diopsys Electrodes. Next, subjects will receive the FL Flicker test three times using the Diopsys device and Diopsys Electrodes.
  Interventions: Diagnostic Test: Electroretinography
- Diopsys device with LKC Electrode Arrays (Other): Subjects will receive the PhNR test three times using the Diopsys device with LKC Electrode Arrays, followed by the FL Flicker test three times using the Diopsys device with the LKC electrode arrays.
  Interventions: Diagnostic Test: Electroretinography
- LKC device with the LKC electrode arrays (Other): Subjects will receive the PhNR test three times using the LKC device with the LKC electrode arrays, followed by the FL Flicker test three times using the LKC device with the LKC electrode arrays.
  Interventions: Diagnostic Test: Electroretinography

INTERVENTIONS:
Diagnostic Test: Electroretinography — Two different electroretinogram devices (Diopsys NOVA and LKC RETeval Devices) will be evaluated with two different electrode arrays (Diopsys Lid Electrodes and LKC RETeval Self-Adhering Electrode Arrays).
  Other Names: Electrode Arrays

SUMMARY:
To compare the Diopsys NOVA and LKC RETeval Devices using the Diopsys Lid Electrodes and LKC RETeval Self-Adhering Electrode Arrays.

DETAILED DESCRIPTION:
This study is an open label, prospective study comparing the Diopsys NOVA and LKC RETeval devices using the Diopsys Lid Electrodes and the LKC RETeval Self-Adhering Electrode Arrays.

Subjects will receive the PhNR test three times using the Diopsys device and Diopsys Electrodes. Next, subjects will receive the FL Flicker test three times using the Diopsys device and Diopsys Electrodes. There will be a short break (10 to 15 minutes), then subjects will receive the PhNR test three times using the Diopsys device with LKC Electrode Arrays, followed by the FL Flicker test three times using the Diopsys device with the LKC electrode arrays. Subjects will receive another short break (5 to 10 minutes), then receive the PhNR test three times using the LKC device with the LKC electrode arrays, followed by the FL Flicker test three times using the LKC device with the LKC electrode arrays.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 22 years of age on day of enrollment
* BCVA letter score of 75 or better (Snellen equivalent of 20/32 or better) on day of enrollment
* Eyes are healthy/normal based on prior examinations, record review, and/or patient intake questions. Subject has not been diagnosed with any ocular pathology that could affect ERG results.
* Able to communicate well with the Investigator and able to understand and comply with the requirements of the study
* Informed of the nature of this study and has provided written, informed consent in accordance with institutional, local and national regulatory guidelines

Exclusion Criteria:

* A spherical refraction outside + 5.0 D and cylinder correction outside + 3.0 D on day of enrollment
* Intraocular surgery (except non-complicated cataract or refractive surgery performed more than 1 year before enrollment)
* Any prior macular or panretinal photocoagulation laser treatment
* History of ophthalmic or neurologic condition known to affect visual function
* Inability to obtain a reliable ERG test
* History of Diabetic retinopathy
* History of Glaucoma
* History of ARMD
* History of seizure disorder
* Has an open sore(s) or dermatological condition that may come in contact with the electrodes/electrode arrays
* In the opinion of the Investigator, is unlikely to comply with the study protocol

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
PhNR Latency (ms) | Day 1
  Change in ERG PhNR Latency (ms) parameter

SECONDARY OUTCOMES:
FL Latency (ms) | Day 1
  Change in ERG FL Latency (ms) parameter

OTHER OUTCOMES:
PhNR B-wave Latency (ms) | Day 1
  Change in ERG PhNR B-wave Latency (ms) parameter
FL Magnitude (µV) | Day 1
  Change in ERG FL Magnitude (µV) parameter
PhNR A-Wave Latency (ms) | Day 1
  Change in ERG PhNR A-Wave Latency (ms) parameter
PhNR Ratio | Day 1
  Change in ERG PhNR Ratio parameter
PhNR amplitude (µV) | Day 1
  Change in ERG PhNR amplitude (µV) parameter
PhNR B-Wave Amplitude (µV) | Day 1
  Change in ERG PhNR B-Wave Amplitude (µV) parameter
PhNR A-Wave Amplitude (µV) | Day 1
  Change in ERG PhNR A-Wave Amplitude (µV) parameter
FL Phase (deg) | Day 1
  Change in ERG FL Phase (deg) parameter

CONTACTS AND LOCATIONS:
Overall Officials: Nate Lighthizer, OD, Principal Investigator — NSU Oklahoma College of Optometry
Locations (1):
- NSU Oklahoma College of Optometry, Tahlequah, Oklahoma, United States